CLINICAL TRIAL: NCT03903172
Title: Post-partum Non-pharmacologic Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wright State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06605
Record Dates: First submitted 2019-03-15; First posted 2019-04-04 (Actual); Results first posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-03

CONDITIONS: Pain Management; Vaginal Delivery
Keywords: pain management; vaginal delivery; nonpharmacologic; abdominal binder
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Non-blinded, parallel group
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Binder Arm (Experimental): Abdominal binder + standard of care postpartum pain management
  Interventions: Device: Abdominal binder
- Standard of Care (No Intervention): Standard of care postpartum pain managment

INTERVENTIONS:
Device: Abdominal binder — Abdominal binder
  Arms: Binder Arm

SUMMARY:
This study aims to examine whether use of an abdominal binder for postpartum patients after vaginal delivery can effectively manage their pain and reduce the need for pharmacologic analgesics. The investigators hypothesize that use of an abdominal binder will decrease patient pain as reported on a visual analog scale of one to ten, and will decrease quantity of pain medications given. The study will be conducted at the Berry Women's Center at Miami Valley Hospital. Potential eligible participants will be approached regarding the study on admission to labor and delivery. The investigators will recruit 130 participants that will be randomized to two study arms, standard care and standard care plus abdominal binder with 65 participants in each study arm. Data will be collected prospectively while participants are admitted, and through review of electronic medical records. Potential benefits of this study include investigation of a cost-effective method for pain management that could improve patient comfort and reduce need for medications.

DETAILED DESCRIPTION:
Hypothesis Use of an abdominal binder postpartum after a vaginal delivery will be associated with lower pain scores and reduced need for pharmacologic analgesics.

Background A significant part of postpartum care involves management of patients' pain and discomfort. Etiologies of this pain include perineal pain, incisional pain, uterine involution pain, and pelvic girdle and lower back pain. Postpartum pain management primarily focuses on the former three types of pain: perineal, incisional and uterine involution. In a review of the management of postpartum pain, Eshkevari et al discuss several well-established pain management strategies employed for postpartum patients, including ibuprofen and other NSAIDs for uterine involution pain and inflammation; local anesthetics for perineal lacerations or episiotomies; warm or cold compresses for perineal pain; and opioids for post-operative or poorly controlled postpartum pain.

Data regarding management of pelvic girdle and lower back pain is scarce and the limited literature available primarily focus on the pregnant patient. Different proposed treatment or management strategies during pregnancy include physical therapy, targeted exercises, acupuncture, NSAIDS and opioids. Approximately 25% of postpartum women endorse pelvic girdle and/or lower back pain, and these types of pain can persist for as long as several weeks to 1-2 years after delivery. Therefore, management remains key for the postpartum patient as well. The proposed pathophysiology behind pelvic girdle pain and lower back pain in the context of pregnancy is widening of the pubic symphysis and increased laxity in the sacro-iliac joints (SIJ) secondary to both biomechanical shear forces of increased weight bearing and elevated levels of relaxin, a polypeptide hormone that increase laxity of ligaments. A prospective study investigating the impact of abdomino-pelvic belts at different positions on the laxity of the SIJ found that use of the abdomino-pelvic belt significantly decreased mobility of the SIJ. Additionally, pelvic belts or abdominal binders may help provide stability to muscles of the abdomen, back and spine.

Studies investigating the use of abdominal binders for pain management in post-operative patients following both cesarean section and gynecologic surgery have had mixed results. A randomized control trial examining impact of abdominal binders on patient reported pain and symptom distress found no significant difference in pain on post-operative days one and two, and the difference in distress on post-operative day two was no longer statistically significant after correction for multiple measures. Another study involving gynecologic surgery patients randomized to abdominal binder or control groups found that there was no overall significant difference in morphine use or pain scale between the groups, and the benefits were limited to a significant effect on post-operative ambulation for a subset of patients with highest risk of complications: patients > 50 years, cancer patients, and those with vertical incision. In contrast, a more recent randomized controlled trial assessing abdominal binders following cesarean delivery found that pain and symptom distress scores were significantly lower at all time points in comparison to a control group.

A common theme in the current literature regarding postpartum pain management is the need for more research. In light of the current opioid abuse epidemic, which affects approximately 2.1 million people and the U.S Department of Health and Human Services declared a public health emergency in 2017, there is a renewed emphasis utilizing non-opioid methods on pain control. As a primary source of pain in the postpartum period is associated with musculoskeletal pelvic discomfort, the use of a supportive abdomino-pelvic belt may be a non-pharmacologic modality that could reduce pain and decrease narcotic requirements in postpartum patients. No studies have directly assessed the effectiveness of abdominal binders on pain management in postpartum patients. This study aims to examine how use of an abdominal binder might impact postpartum pain, and the use of pharmacologic analgesia following vaginal delivery.

Protocol

* Recruitment

  o Patients admitted to Labor and Delivery will be evaluated for potential participation in the study based on the inclusion and exclusion criteria outlined below. If appropriate to approach, eligible potential participants will be approached in their labor and delivery room prior to delivery. If interested in participation, the Informed Consent document will be presented and explained in the room to ensure privacy.
* Subject Informed Consent

  * Informed consent process will take place at the Berry Women's Center at Miami Valley Hospital
  * Written and signed consent will be obtained in English.
* Plans of obtaining informed consent:

  o Potential eligible participants will be approached in the labor and delivery room to ensure privacy. The research assistant will provide and discuss an informed consent form with the participant. The informed consent form will describe the project goals, length and rational, as well as the types of PHI that will be collected. All participants who agree to participate in the study will sign the informed consent form. All participants will be provided with a copy of the signed consent form.
* Study design and procedures

  * After signing informed consent, participants will be assigned to the intervention or control group via block randomization
  * Those participants in the standard of care group will receive routine postpartum care
  * Those participants in the intervention group will receive an abdominal binder in addition to routine postpartum care
  * Determination of appropriate binder size will be based on a visual assessment of the patient's abdominal circumference
  * Nursing staff will evaluate participant's pain level using a visual analog scale of 1-10 a minimum of every 4 hours. Patient reported pain score and pain location will be recorded in the participant's electronic medical record. These processes do not deviate from current standards of care and documentation.
  * Additional non-pharmacologic pain relief measures utilized by patients will be documented on the data collection sheet attached to the patient's chart. These measures include heating pad, ice pack, and tucks pads
  * All medications received will be documented in the electronic medical record per usual documentation protocols
* Sample Size Estimation & Data Analysis Plan

  * Sample size was estimated using G*Power. In order to detect a difference between groups on pain scores and use of pain medications, 65 patients per group will need to be enrolled. This will enable the investigators to detect a moderate difference (i.e., medium effect size) between the groups with a power = 80% and p at <0.05.
  * The two groups will be compared for 1. reported pain scores (assessed by nursing staff and documented in the EMR) and for 2. pain medications used (morphine equivalent as recorded in the MAR) for the duration of patients' hospital stay. T-test will be used to compare the groups on average pain scores and total pain medication use. Repeated measures analysis of variance will be used to determine differences between the groups over time.
* Data collection plan

  * Prospective data collection with hard copy data entry form that includes PHI for participant identification, basic demographic information, delivery information (see separate document), non-pharmacologic pain relief measures used
  * Electronic medical record review for: pain scores, pain location, medications received
  * Pain score immediately postpartum
  * Pain scores (average scores) on PPD#0 and PPD#1
  * Patient reported pain locations
  * Quantity (total) of non-narcotic pain medication received on PPD#0 and PPD#1
  * Quantity (total) of narcotic pain medication received on PPD#0 and PPD#1
* Risks

  * Allergic reaction to fabric of abdominal binder
  * Skin irritation
  * Increased discomfort or pain with use of abdominal binder
* Mitigation of risks o If participants experience an allergic reaction or skin irritation from the abdominal binder symptomatic treatment will be offered. Participants in the experimental arm will be encouraged to keep the abdominal binders in place for 24 hours postpartum, but will be permitted to remove the abdominal binder at any time should it cause irritation, increased pain or any other adverse reaction.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Pregnant
* Admitted to labor and delivery
* Anticipated spontaneous vaginal delivery
* Informed consent obtained

Exclusion Criteria:

* Documented chronic pain condition
* Chronic narcotic use or Maternal Abstinence Treatment
* UDS positive for opiates on admission
* Trial of labor after cesarean
* Lack of sufficient English proficiency to obtain informed consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women will be enrolled
Enrollment: 105 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheela Barhan, MD, Principal Investigator — Wright State University
Locations (1):
- Miami Valley Hospital, Dayton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shard on a case by case basis.

REFERENCES:
- [Background] Eshkevari L, Trout KK, Damore J. Management of postpartum pain. J Midwifery Womens Health. 2013 Nov-Dec;58(6):622-31. doi: 10.1111/jmwh.12129. PMID 24406035
- [Background] Wu WH, Meijer OG, Uegaki K, Mens JM, van Dieen JH, Wuisman PI, Ostgaard HC. Pregnancy-related pelvic girdle pain (PPP), I: Terminology, clinical presentation, and prevalence. Eur Spine J. 2004 Nov;13(7):575-89. doi: 10.1007/s00586-003-0615-y. Epub 2004 Aug 27. PMID 15338362
- [Background] Vermani E, Mittal R, Weeks A. Pelvic girdle pain and low back pain in pregnancy: a review. Pain Pract. 2010 Jan-Feb;10(1):60-71. doi: 10.1111/j.1533-2500.2009.00327.x. Epub 2010 Oct 26. PMID 19863747
- [Background] Mens JM, Damen L, Snijders CJ, Stam HJ. The mechanical effect of a pelvic belt in patients with pregnancy-related pelvic pain. Clin Biomech (Bristol). 2006 Feb;21(2):122-7. doi: 10.1016/j.clinbiomech.2005.08.016. Epub 2005 Oct 7. PMID 16214275
- [Background] Liddle SD, Pennick V. Interventions for preventing and treating low-back and pelvic pain during pregnancy. Cochrane Database Syst Rev. 2015 Sep 30;2015(9):CD001139. doi: 10.1002/14651858.CD001139.pub4. PMID 26422811
- [Background] Gillier CM, Sparks JR, Kriner R, Anasti JN. A randomized controlled trial of abdominal binders for the management of postoperative pain and distress after cesarean delivery. Int J Gynaecol Obstet. 2016 May;133(2):188-91. doi: 10.1016/j.ijgo.2015.08.026. Epub 2016 Jan 14. PMID 26892694
- [Background] Ghana S, Hakimi S, Mirghafourvand M, Abbasalizadeh F, Behnampour N. Randomized controlled trial of abdominal binders for postoperative pain, distress, and blood loss after cesarean delivery. Int J Gynaecol Obstet. 2017 Jun;137(3):271-276. doi: 10.1002/ijgo.12134. Epub 2017 Mar 28. PMID 28241386
- [Derived] Deussen AR, Ashwood P, Martis R, Stewart F, Grzeskowiak LE. Relief of pain due to uterine cramping/involution after birth. Cochrane Database Syst Rev. 2020 Oct 20;10(10):CD004908. doi: 10.1002/14651858.CD004908.pub3. PMID 33078388

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Binder Arm | Standard of Care
Started | 54 | 51
Completed | 50 | 50
Not Completed | 4 | 1
Not completed — screen fail | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Binder Arm | Standard of Care | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.4 (6.0) | 23.2 (3.9) | 24.8 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100
Postpartum pain score (standard scale is 0 - no pain to 10- severe pain) [Mean (Standard Deviation); unit: units on a scale] — First pain score after delivery
  units on a scale | 0.68 (1.68) | 0.16 (0.65) | 0.42 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Patient Reported Average Pain Score
Description: Pain score (standard scale is 0 - no pain to 10- severe pain) will be recorded by nursing staff in electronic medical record per standard of care. Average pain score for postpartum day 0 and postpartum day 1 will be computed. High scores represent greater pain.
Time Frame: Average score computed from postpartum day 0, postpartum day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Binder Arm | Standard of Care
Number analyzed (Participants) | 50 | 50
units on a scale
  Average pain on postpartum Day 0 | 1.37 (1.35) | 1.06 (1.60)
  Average pain on postpartum Day 1 | 2.03 (1.6) | 2.41 (1.3)
Statistical Analysis 1: Comparison: Binder Arm vs Standard of Care; Day 0; Test type: Superiority; p = 0.25, t-test, 2 sided
Statistical Analysis 2: Comparison: Binder Arm vs Standard of Care; Day 1; Test type: Superiority; p = .93, t-test, 2 sided

2. Primary Outcome: Number of Patient Using Each Type of Non-narcotic Pain Medications
Description: Number of patients using each type of non-narcotic pain medication as recorded on MAR for postpartum day 0 and postpartum day 1
Time Frame: Number of patients using each type of non-narcotic medication recorded on postpartum day 0 and postpartum day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Binder Arm | Standard of Care
Number analyzed (Participants) | 50 | 50
Participants
  Acetaminophen | 30 | 30
  Ibuprofen | 1 | 2
  Cyclobenzaprine | 1 | 2
  Methocarbamol | 1 | 6
  Hydroxyzine | 0 | 2
  Other | 6 | 5
Statistical Analysis 1: Comparison: Binder Arm vs Standard of Care; Used acetominophen; Test type: Superiority; p = 1.0, Fisher Exact
Statistical Analysis 2: Comparison: Binder Arm vs Standard of Care; Used ibuprofen; Test type: Superiority; p = 1.0, Fisher Exact
Statistical Analysis 3: Comparison: Binder Arm vs Standard of Care; Used Cyclobenzaprine; Test type: Superiority; p = 1.0, Fisher Exact
Statistical Analysis 4: Comparison: Binder Arm vs Standard of Care; Used Methocarbamol; Test type: Superiority; p = .11, Fisher Exact
Statistical Analysis 5: Comparison: Binder Arm vs Standard of Care; Used Hydroxyzine; Test type: Superiority; p = .49, Fisher Exact
Statistical Analysis 6: Comparison: Binder Arm vs Standard of Care; Used an 'Other' non-pharmacologic medication; Test type: Superiority; p = 1.0, Fisher Exact

3. Primary Outcome: Any Narcotic Pain Medication Use
Description: Any narcotic pain medication use (yes/no) as recorded on MAR for postpartum day 0 and postpartum day 1
Time Frame: Any narcotic medication use from postpartum day 0 and postpartum day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Binder Arm | Standard of Care
Number analyzed (Participants) | 50 | 50
Participants | 4 | 2
Statistical Analysis 1: Comparison: Binder Arm vs Standard of Care; Any narcotic medication used; Test type: Superiority; p = 1.0, Fisher Exact

ADVERSE EVENTS:
Time Frame: After delivery (postpartum Day 0) to hospital discharge (postpartum Day 1)
Description: This is a low risk population
Arm/Group | Binder Arm | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

LIMITATIONS AND CAVEATS:
While the initial sample size estimate indicated a requirement of 64 patients per group, the effect size was much smaller than anticipated, limiting the overall study power and the ability to detect a difference. This study was unblinded for the medical team and patients. It was not possible to determine the total length of time patients were wearing the abdominal binders. Binders were applied within the first two hours postpartum, and documented in the EMR, removal was not always documented.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/72/NCT03903172/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/72/NCT03903172/SAP_001.pdf